CLINICAL TRIAL: NCT02775903
Title: A Randomized, Multicenter, Open-label, Phase 2 Study Evaluating the Efficacy and Safety of Azacitidine Subcutaneous in Combination With Durvalumab (MEDI4736) in Previously Untreated Subjects With Higher-Risk Myelodysplastic Syndromes (MDS) or in Elderly (>= 65 Years) Acute Myeloid Leukemia (AML) Subjects Not Eligible for Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: An Efficacy and Safety Study of Azacitidine Subcutaneous in Combination With Durvalumab (MEDI4736) in Previously Untreated Adults With Higher-Risk Myelodysplastic Syndromes (MDS) or in Elderly Patients With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-MDS-001
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes
Keywords: MEDI4736; Durvalumab; Myelodysplastic Syndromes; Acute Myeloid Leukemia; Hematopoietic Stem Cell Transplantation; Azacitidine; Safety; Efficacy; PD-L1
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azacitidine + Durvalumab (Experimental): Participants received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks (Q4W) in combination with 1500 mg intravenous durvalumab on Day 1 of every 4 week cycle for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
  Interventions: Drug: Azacitidine; Biological: Durvalumab
- Azacitidine Alone (Active Comparator): Participants received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Administered by subcutaneous injection on Days 1 to 7 of each 4-week treatment cycle.
Biological: Durvalumab — Administered by intravenous infusion on Day 1 of every 4-week treatment cycle.
  Other Names: MEDI4736
  Arms: Azacitidine + Durvalumab

SUMMARY:
The primary objective of this study is to evaluate the efficacy of subcutaneous azacitidine in combination with durvalumab as compared with subcutaneous azacitidine alone in adults with previously untreated, higher risk MDS who are not eligible for HSCT or in adults ≥ 65 years old with previously untreated AML who are not eligible for HSCT, with intermediate or poor cytogenetic risk.

ELIGIBILITY:
Inclusion Criteria:

For both cohorts:

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Female subjects of childbearing potential may participate, providing they meet the following conditions:

   1. Have 2 negative pregnancy tests as verified by the Investigator prior to starting any investigational product (IP) therapy: serum pregnancy test at screening and negative serum or urine pregnancy test (Investigator's discretion) within 72 hours prior to starting treatment with IP (Cycle 1, Day 1). They must agree to ongoing pregnancy testing during the course of the study (before beginning each subsequent cycle of treatment), and after the last dose of any IP. This applies even if the subject practices complete abstinence from heterosexual contact.
   2. Agree to practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to the use of a highly effective method of contraception use from 28 days prior to starting durvalumab or azacitidine, and must agree to continue using such precautions while taking durvalumab or azacitidine (including dose interruptions) and up to 90 days after the last dose of durvalumab or azacitidine. Cessation of contraception after this point should be discussed with a responsible physician.
   3. Agree to abstain from breastfeeding during study participation and for at least 90 days after the last dose of IP.
   4. Refrain from egg cell donation while taking durvalumab and for at least 90 days after the last dose of durvalumab.
4. Male subject must:

   1. Either practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to avoid fathering a child, to use highly effective methods of contraception, male condom plus spermicide during sexual contact with a pregnant female or a female of childbearing potential (even if he has undergone a successful vasectomy) from starting dose of IP (Cycle 1 Day 1), including dose interruptions through 90 days after receipt of the last dose of durvalumab or azacitidine.
   2. Refrain from semen or sperm donation while taking IP and for at least 90 days after the last dose of IP.
5. Understand and voluntarily sign a biomarker-specific component of the informed consent form prior to any study-related procedures conducted.
6. Willing and able to adhere to the study visit schedule and other protocol requirements.

   MDS Cohort:
7. Age ≥ 18 years at the time of signing the informed consent form.
8. Central confirmation of diagnosis of previously untreated primary or secondary myelodysplastic syndromes (MDS) as per World Health Organization (WHO) classification. Results of central pathology review are required prior to receiving the first dose of IP.
9. Central confirmation of the categorization of the MDS risk classification, as per the Revised - International prognostic scoring system (IPSS-R) Intermediate risk with >10% blasts or poor or very poor cytogenetics, or IPSS-R High or Very High risk (results of central pathology review required prior to receiving the first dose of IP).

   Acute myeloid leukemia (AML) Cohort:
10. Age ≥ 65 years at the time of signing the informed consent form (ICF).
11. Central confirmation of diagnosis of one of the following untreated AML as per WHO classification:

    * Newly diagnosed, histologically confirmed de novo AML (bone marrow blasts ≥ 20%), or
    * AML secondary to prior MDS, or
    * AML secondary to exposure to potentially leukemogenic therapies or agents (eg, radiation therapy, alkylating agents, topoisomerase II inhibitors) with the primary malignancy in remission for at least 2 years.
12. Central confirmation of intermediate or poor risk status, based on Cytogenetics for acute myeloid leukemia.

Exclusion Criteria:

For both cohorts:

1. Prior hematopoietic stem cell transplant.
2. Considered eligible for hematopoietic stem cell transplant (allogeneic or autologous) at the time of signing the ICF.
3. Prior exposure to azacitidine, decitabine or prior exposure to the investigational oral formulation of decitabine, or other oral azacitidine derivative.
4. Inaspirable bone marrow.
5. Use of any of the following within 28 days prior to the first dose of IP:

   * Thrombopoiesis-stimulating agents (eg, romiplostim, eltrombopag, Interleukin-11)
   * Any hematopoietic growth factors (erythropoietin-stimulating agents [ESAs], granulocyte colony-stimulating factor (G-CSF) and other red blood cell (RBC) hematopoietic growth factors (eg, Interleukin-3)
   * Any investigational agents within 28 days or 5 half-lives (whichever is longer) of initiating study treatment
6. Prior history of malignancies (except MDS for AML subjects), unless the subject has been free of the disease for ≥ 2 years. However, subjects with the following history/concurrent conditions are allowed:

   * Basal or squamous cell carcinoma of the skin
   * Carcinoma in situ of the cervix
   * Carcinoma in situ of the breast
   * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [tumor, node, metastases (TNM)] clinical staging system).
7. Pregnant or breast-feeding females or females who intend to become pregnant during study participation.
8. Subject has active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis with the exception of a prior episode that has resolved or diverticulosis, celiac disease, irritable bowel disease [exclude only if active within the last 6 months prior to signing the ICF], or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener's syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis; etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

   * Subjects with vitiligo or alopecia;
   * Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement for ≥ 3 months prior to signing the ICF; or
   * Subjects with psoriasis not requiring systemic treatment
9. Significant active cardiac disease within the previous 6 months prior to signing the ICF, including:

   * New York Heart Association (NYHA) Class III or IV congestive heart failure;
   * Unstable angina or angina requiring surgical or medical intervention; and/or
   * Significant cardiac arrhythmia
   * Myocardial infarction
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment), uncontrolled hypertension, cardiac arrhythmia, pneumonitis, interstitial lung disease, active peptic ulcer disease or gastritis that would limit compliance with study requirement.
11. Known human immunodeficiency virus (HIV) or hepatitis C (HCV) infection, or evidence of active hepatitis B virus (HBV) infection.
12. Known or suspected hypersensitivity to azacitidine, mannitol, or durvalumab, its constituents, or to any other humanized monoclonal antibody.
13. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
14. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
15. Prior anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), programmed death-1 (PD-1), or programmed death ligand-1 (PD-L1) or other immune checkpoint mAb exposure.
16. Other investigational monoclonal antibodies (mAbs) within 6 months prior to first dose of IP.
17. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of IP. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical, or local steroid injections (eg, intra-articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication)
18. History of primary immunodeficiency.
19. Receipt of live, attenuated vaccine within 30 days prior to the first dose of IP (NOTE: Subjects, if enrolled, should not receive live vaccine during the study and for 30 days after the last dose of durvalumab).
20. Unwilling or unable to complete subject reported outcome assessments without assistance or with minimal assistance from trained site personnel and/or caregiver.
21. Subjects who have had clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS leukemia.
22. Presence of advanced malignant hepatic tumors.
23. Any of the following laboratory abnormalities:

    * Serum aspartate aminotransferase (AST/SGOT) or alanine aminotransferase (ALT/SGPT) > 2.5 × upper limit of normal (ULN)
    * Serum total bilirubin > 1.5 × ULN. Higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis). Subjects are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Coombs' test or over 50% of indirect bilirubin
    * Serum creatinine > 2.5 × ULN.

    MDS Cohort:
24. Any previous cytotoxic, cytostatic, hormonal, biological or immunological treatment for MDS (ESA with or without G-CSF are allowed under certain conditions, see exclusion criterion # 5).
25. Any investigational therapy within 28 days prior to the first dose of IP.
26. Use of hydroxyurea within 2 weeks prior to obtaining the screening hematology sample and prior to first dose of IP.
27. Absolute white blood cell (WBC) count ≥ 15 × 10^9/L.

    AML Cohort:
28. Previous cytotoxic, cytostatic, hormonal, biological or immunological treatment (ESA with or without G-CSF and iron chelating therapy and hydroxyurea are allowed under certain conditions, see exclusion criterion #5) or biologic treatment for AML.
29. Any investigational therapy within 28 days prior to the first dose of IP.
30. Use of hydroxyurea within 2 weeks prior to obtaining the screening hematology sample and prior to first dose of IP.
31. Prior use of targeted therapy agents (eg, FLT3 inhibitors, other kinase inhibitors).
32. Suspected or proven acute promyelocytic leukemia (French-American-British (FAB) M3) based on morphology, immunophenotype, molecular assay, or karyotype; AML associated with t(9;22) karyotype, biphenotypic acute leukemia or AML with previous hematologic disorder such as chronic myelogenous leukemia or myeloproliferative neoplasms.
33. Acute myeloid leukemia associated with inv(16), t(8;21), t(16;16), t(15;17) karyotypes or molecular evidence of such translocations if not associated with a c-Kit mutation.
34. Absolute WBC count ≥ 15 × 10^⁹/L (NOTE: Hydroxyurea is not allowed to attain a WBC count ≤ 15 x 10⁹/L).
35. Known history or presence of Sweet Syndrome at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CL Beach, Pharm D, Study Director — Celgene Corporation
Locations (103):
- United States (12):
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas- MD Anderson, Houston, Texas
- Austria (7):
  - Medizinische Universitat Graz, Graz
  - Medizinische Universitat Innsbruck, Innsbruck
  - Elisabethinen Hospital Linz, Linz
  - Salzburger Landkliniken St. Johanns-Spital, Salzburg
  - Hanusch Krankenhaus der Stadt Wien, Vienna
  - Local Institution - 653, Vienna
  - AKH Wien, Wein
- Belgium (6):
  - Cliniques Universitaires St-Luc, Brussels
  - Grand Hopital de Charleroi, Charleroi
  - Local Institution - 202, Ghent
  - UH Gent, Ghent
  - UH Gasthuisberg, Leuven
  - Cliniques Universitaires UCL de Mont-Godine, Yvoir
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Ottawa General Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM - Notre Dame, Montreal, Quebec
- France (13):
  - Centre Hospitalier Universitaire d' Angers, Angers
  - Hopital Avicenne, Bobigny
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire de Grenoble Hopital Albert Michallon, La Tronche
  - Centre Leon Berard, Lyon
  - Local Institution - 261, Lyon
  - CHRU de Nantes - Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Local Institution - 251, Paris
  - CHU Bordeaux, Pessac
  - Local Institution - 254, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - IUCT Oncopole, Toulouse
- Germany (13):
  - Local Institution - 604, Dresden
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Local Institution - 603, Düsseldorf
  - Marien Hospital, Düsseldorf
  - Universitatsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe Universitat, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule HannoverZentrum Innere Medizin, Hanover
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum der LMU Campus Grosshadern, München
  - Local Institution - 605, München
  - Klinikum rechts der Isar der TU Munchen, München
  - Universitatsklinikum Ulm, Ulm
- Italy (13):
  - AO Spedali Civili di Brescia, Brecia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Niguarda Milano, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - I.R.C.C.S. Policlinico San Matteo - Universita di Pavia, Pavia
  - Local Institution - 302, Pavia
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Roma
  - Local Institution - 303, Roma
  - Policlinico Agostino Gemelli - Istituto di Ematologia, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Local Institution - 304, Rome
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia die Udine, Udine
  - Universita degli Studi dell'Insubria - Ospedale di Circolo e Fondazione Macchi - Varese, Varese
- VU University Medical Center, Amsterdam, Netherlands
- Poland (5):
  - Oddzial Hematologii Onkologicznej Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologicz, Brzozów
  - Katedra i Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 1 Klinika Hematoonkologii i Transplantacji Szpiku, Lubin
  - Oddzial Hematologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej MSW, Olsztyn
  - Klinika Hematologii Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
- Portugal (5):
  - Hospitais da Universidade de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil EPE, Lisbon
  - Ipo Instituto Portugues De Oncologia Porto, Porto
  - Local Institution - 502, Porto
  - Hospital de Sao Joao, Porto
- Spain (13):
  - Hospital Universitario Vall D hebron, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Complejo Hospitalario San Pedro de Alcantara, Cáceres
  - Hospital Universitario La Princesa, Madrid
  - Hospital Gregorio Maranon, Madrid
  - Local Institution - 555, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario La Fe, Valencia
  - Local Institution - 559, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (9):
  - University Hospital Birmingham, Birmingham
  - St James University Hospital, Leeds
  - St Bartholomews Hospital, London
  - Kings College Hospital, London
  - University College London Hospital, London Bloomsbury
  - The Christie NHS Foundation Trust, Manchester
  - John Radcliffe Hospital, Oxford
  - Local Institution - 453, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Bewersdorf JP, Hasle V, Shallis RM, Thompson E, Lopes de Menezes D, Rose S, Boss I, Mendez L, Podoltsev N, Stahl M, Kewan T, Halene S, Haferlach T, Fox BA, Zeidan AM. Integrated Immune Landscape Analysis of RNA Splicing Factor-Mutant AML and Higher risk MDS Treated with Azacitidine +/- Durvalumab. Ther Adv Hematol. 2025 Jun 21;16:20406207251347344. doi: 10.1177/20406207251347344. eCollection 2025. PMID 40546817
- [Derived] Zeidan AM, Bewersdorf JP, Hasle V, Shallis RM, Thompson E, de Menezes DL, Rose S, Boss I, Halene S, Haferlach T, Fox BA. Integrated genetic, epigenetic, and immune landscape of TP53 mutant AML and higher risk MDS treated with azacitidine. Ther Adv Hematol. 2024 Jun 15;15:20406207241257904. doi: 10.1177/20406207241257904. eCollection 2024. PMID 38883163
- [Derived] Zeidan AM, Boss I, Beach CL, Copeland WB, Thompson E, Fox BA, Hasle VE, Ogasawara K, Cavenagh J, Silverman LR, Voso MT, Hellmann A, Tormo M, O'Connor T, Previtali A, Rose S, Garcia-Manero G. A randomized phase 2 trial of azacitidine with or without durvalumab as first-line therapy for higher-risk myelodysplastic syndromes. Blood Adv. 2022 Apr 12;6(7):2207-2218. doi: 10.1182/bloodadvances.2021005487. PMID 34972214
- [Derived] Zeidan AM, Boss I, Beach CL, Copeland WB, Thompson E, Fox BA, Hasle VE, Hellmann A, Taussig DC, Tormo M, Voso MT, Cavenagh J, O'Connor T, Previtali A, Rose S, Silverman LR. A randomized phase 2 trial of azacitidine with or without durvalumab as first-line therapy for older patients with AML. Blood Adv. 2022 Apr 12;6(7):2219-2229. doi: 10.1182/bloodadvances.2021006138. PMID 34933333
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 cohorts: • Adults with previously untreated intermediate, high or very high risk myelodysplastic syndromes (MDS) not eligible for hematopoietic stem cell transplantation (HSCT). • Adults with previously untreated acute myeloid leukemia (AML) ≥ 65 years and not eligible for HSCT with intermediate or poor cytogenetic risk.
Pre-assignment Details: Within each cohort participants were randomized in a 1:1 ratio to receive either azacitidine plus durvalumab or azacitidine alone. Randomization was stratified according to cytogenetic risk: • Very good, good and intermediate versus poor and very poor for MDS • Intermediate versus poor for AML .
Groups:
- MDS: Azacitidine + Durvalumab: Participants with MDS received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks (Q4W) in combination with 1500 mg intravenous durvalumab on Day 1 of every 4 week cycle for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
- MDS: Azacitidine Alone: Participants with MDS received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
- AML: Azacitidine + Durvalumab: Participants with AML received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks (Q4W) in combination with 1500 mg intravenous durvalumab on Day 1 of every 4 week cycle for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
- AML: Azacitidine Alone: Participants with AML received 75 mg/m² subcutaneous azacitidine for 7 days every 4 weeks for at least 6 cycles. Participants who benefited from treatment may have continued treatment until loss of that benefit, disease progression or other treatment discontinuation criterion were met.
Period: Overall Study
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Started | 42 | 42 | 64 | 65
Completed | 4 | 1 | 1 | 5
Not Completed | 38 | 41 | 63 | 60
Not completed — Death | 7 | 11 | 12 | 11
Not completed — Adverse Event | 0 | 1 | 12 | 3
Not completed — Progressive disease | 15 | 14 | 30 | 20
Not completed — Lack of Efficacy | 2 | 2 | 2 | 6
Not completed — Withdrawal by Subject | 7 | 5 | 5 | 8
Not completed — Other reasons | 7 | 8 | 2 | 12

BASELINE CHARACTERISTICS:
Population: All randomized participants (intent-to-treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone | Total
Number analyzed (Participants) | 42 | 42 | 64 | 65 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were collected and reported separately for each cohort.
  years
    MDS: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS | 72.5 (6.53) | 73.2 (8.83) |  |  | 72.8 (7.72)
    AML: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML |  |  | 76.2 (5.97) | 75.3 (5.36) | 75.8 (5.67)
Age, Customized [Count of Participants; unit: Participants] — Population: Data were collected and reported separately for each cohort.
  Participants
    MDS Cohort: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS Cohort: < 65 years | 2 | 10 |  |  | 12
    MDS Cohort: ≥ 65 to < 75 years | 21 | 11 |  |  | 32
    MDS Cohort: ≥ 75 years | 19 | 21 |  |  | 40
    AML Cohort: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML Cohort: < 65 years |  |  | 0 | 0 | 0
    AML Cohort: ≥ 65 to < 75 years |  |  | 24 | 28 | 52
    AML Cohort: ≥ 75 years |  |  | 40 | 37 | 77
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were collected and reported separately for each cohort.
  Participants
    MDS Cohort: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS Cohort: Female | 14 | 12 |  |  | 26
    MDS Cohort: Male | 28 | 30 |  |  | 58
    AML Cohort: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML Cohort: Female |  |  | 24 | 34 | 58
    AML Cohort: Male |  |  | 40 | 31 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data were collected and reported separately for each cohort.
  Participants
    MDS Cohort: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS Cohort: Hispanic or Latino | 5 | 2 |  |  | 7
    MDS Cohort: Not Hispanic or Latino | 30 | 33 |  |  | 63
    MDS Cohort: Unknown or Not Reported | 7 | 7 |  |  | 14
    AML Cohort: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML Cohort: Hispanic or Latino |  |  | 6 | 3 | 9
    AML Cohort: Not Hispanic or Latino |  |  | 39 | 41 | 80
    AML Cohort: Unknown or Not Reported |  |  | 19 | 21 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data were collected and reported separately for each cohort.
  Participants
    MDS Cohort: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS Cohort: American Indian or Alaska Native | 0 | 0 |  |  | 0
    MDS Cohort: Asian | 2 | 1 |  |  | 3
    MDS Cohort: Black or African American | 1 | 0 |  |  | 1
    MDS Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    MDS Cohort: White | 30 | 33 |  |  | 63
    MDS Cohort: Not Collected or Reported | 7 | 5 |  |  | 12
    MDS Cohort: Other | 2 | 3 |  |  | 5
    AML Cohort: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML Cohort: American Indian or Alaska Native |  |  | 0 | 0 | 0
    AML Cohort: Asian |  |  | 0 | 0 | 0
    AML Cohort: Black or African American |  |  | 0 | 1 | 1
    AML Cohort: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    AML Cohort: White |  |  | 45 | 42 | 87
    AML Cohort: Not Collected or Reported |  |  | 18 | 21 | 39
    AML Cohort: Other |  |  | 1 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: - 0 = Fully active, no restrictions; - 1 = Restricted activity but ambulatory, able to carry out work of a light nature; - 2 = Ambulatory and capable of all self-care but unable to carry out work activities; - 3 = Limited self-care, confined to bed or chair more than 50% of waking hours; - 4 = Completely disabled, no selfcare, confined to bed or chair; - 5 = Dead Population: Data were collected and reported separately for each cohort.
  Participants
    MDS Cohort: number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    MDS Cohort: 0 - Fully active | 17 | 18 |  |  | 35
    MDS Cohort: 1 - Restricted but ambulatory | 20 | 20 |  |  | 40
    MDS Cohort: 2 - Ambulatory but unable to work | 3 | 4 |  |  | 7
    MDS Cohort: 3 - Limited self-care | 0 | 0 |  |  | 0
    MDS Cohort: 4 - Completely Disabled | 0 | 0 |  |  | 0
    MDS Cohort: Missing | 2 | 0 |  |  | 2
    AML Cohort: number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    AML Cohort: 0 - Fully active |  |  | 19 | 26 | 45
    AML Cohort: 1 - Restricted but ambulatory |  |  | 40 | 32 | 72
    AML Cohort: 2 - Ambulatory but unable to work |  |  | 5 | 7 | 12
    AML Cohort: 3 - Limited self-care |  |  | 0 | 0 | 0
    AML Cohort: 4 - Completely Disabled |  |  | 0 | 0 | 0
    AML Cohort: Missing |  |  | 0 | 0 | 0
Revised International Prognostic Scoring System (IPSS-R) Cytogenetic Risk Groups (MDS Cohort) [Count of Participants; unit: Participants] — The IPSS-R cytogenetic risk score is based on cytogenetic (chromosomal) abnormalities observed in the bone marrow cells. A good cytogenetic prognosis predicts longer survival and lower transformation to leukemia. Population: Participants in the MDS cohort only
  Participants
    number analyzed (Participants) | 42 | 42 | 0 | 0 | 84
    Very good | 1 | 1 |  |  | 2
    Good | 10 | 10 |  |  | 20
    Intermediate | 9 | 8 |  |  | 17
    Poor | 8 | 9 |  |  | 17
    Very Poor | 14 | 14 |  |  | 28
Cytogenetic Risk Classifications (AML Cohort) [Count of Participants; unit: Participants] — Cytogenetic risk classification according to the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology for Acute Myeloid Leukemia. Risk categories are based on analysis of cytogenetics (the study of chromosomes), including chromosomal deletions, duplications, or substitutions and analysis of molecular abnormalities such as specific mutations. Better risk indicates disease more likely to respond to initial treatment and less likely to relapse whereas poor-risk is characterized by poor response to induction chemotherapy and higher relapse rates. Population: Participants in the AML cohort only
  Participants
    number analyzed (Participants) | 0 | 0 | 64 | 65 | 129
    Better risk |  |  | 0 | 0 | 0
    Intermediate risk |  |  | 25 | 26 | 51
    Poor risk |  |  | 16 | 16 | 32
    Missing |  |  | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: MDS Cohort: Overall Response Rate
Description: Overall response rate (ORR) is defined as the percentage of participants achieving a complete remission (CR), partial remission (PR), marrow complete remission (mCR), and/or hematological improvement (HI) based on International Working Group (IWG) 2006 response criteria for MDS and central review. CR: ≤ 5% myeloblasts in bone marrow (BM), and peripheral blood: hemoglobin ≥ 11 g/dL; platelets ≥ 100 × 10⁹/L; neutrophils ≥ 1.0 × 10⁹/L; blasts 0% PR: BM blasts decreased by ≥ 50% but still > 5%; peripheral blood as for CR mCR: BM ≤ 5% myeloblasts and decrease by ≥ 50% HI: Any of the following: •Hemoglobin increase by ≥ 1.5 g/dL or reduction of units of red blood cell (RBC) transfusions of at least 4 RBC transfusions/8 weeks compared with pretreatment •Absolute increase in platelets of ≥ 30 × 10⁹/L if pretreatment value > 20 × 10⁹/L or increase from < 20 × 10⁹/L to > 20 × 10⁹/L and by at least 100% •At least 100% increase in neutrophils and an absolute increase of > 0.5 × 10⁹/L
Time Frame: Response was assessed following every 3 treatment cycles until treatment discontinuation; median duration of treatment was 239 days (AZA) and 215 days (DUR) in the AZA + DUR group and 210 days in the AZA alone group.
Population: All randomized participants in the MDS cohort; participants who discontinued before 6 cycles of treatment without achieving overall response were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 42 | 42
percentage of participants | 61.9 [47.22 to 76.59] | 47.6 [32.51 to 62.72]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Superiority; p = 0.1838, Wald asymptotic two-sided test

2. Primary Outcome: AML Cohort: Overall Response Rate
Description: Overall response rate for AML is defined as the percentage of participants achieving an overall response of morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi) based on modified IWG 2003 response criteria for AML and central review. CR: The following conditions must be met: •Absolute neutrophil count (ANC) ≥ 1.0 x10⁹/L •Platelet count ≥ 100 x10⁹/L •The bone marrow should contain less than 5% blast cells; •Auer rods should not be detectable; •No platelet, or whole blood transfusions for 7days prior to the date of the hematology assessment. CRi: Defined as a morphologic complete remission but the ANC count may be < 1.0 x10⁹/L and/or the platelet count may be < 100 x10⁹/L.
Time Frame: Response was assessed following every 3 treatment cycles until treatment discontinuation; median duration of treatment was 198 days (AZA) and 171 days (DUR) in the AZA + DUR group and 203 days in the AZA alone group.
Population: All randomized participants in the AML cohort; participants who discontinued before 6 cycles of treatment without achieving overall response were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 64 | 65
percentage of participants | 31.3 [19.89 to 42.61] | 35.4 [23.76 to 47.01]
Statistical Analysis 1: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Superiority; p = 0.6180, Wald asymptotic two-sided test

3. Secondary Outcome: MDS Cohort: Kaplan Meier Estimate of Time to First Response
Description: Time to first response is defined as the time from randomization to the earliest date any response (complete remission (CR), partial remission (PR), marrow complete remission (mCR), and/or hematological improvement (HI)) based on International Working Group (IWG) 2006 response criteria for MDS and central review. Participants who did not achieve any defined response were censored at the date of last adequate response assessment, disease progression, or death, whichever occurred first. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization to the earliest date any response (up to approximately 34 months)
Population: All participants randomized in the MDS cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 42 | 42
Weeks | 14.3 [11.3 to 20.9] | 18.4 [8.1 to 26.1]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.7016, Log Rank; Log-rank test stratified according to the cytogenetic risk at time of randomization (very good, good and intermediate vs poor and very poor)

4. Secondary Outcome: MDS Cohort: Kaplan Meier Estimate of Relapse-free Survival
Description: Relapse-free survival is defined as the time from the date of first documented response (complete remission (CR), partial remission (PR)) to the date of disease relapse or death from any cause, whichever occurred first according to the International Working Group (IWG) 2006 response criteria for MDS and central review. Participants who were still alive and progression-free were censored at the date of their last response assessment. Participants who received a subsequent therapy before the date of disease relapse or death were censored at the time of subsequent therapy. Relapse after CR or PR is defined as at least one of the following: •Return to pretreatment bone marrow blast % •Decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets •Reduction in hemoglobin concentration by ≥ 1.5 g/dL or transfusion dependence. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization to to the date of disease relapse or death from any cause, whichever occurred first (up to approximately 34 months)
Population: Participants randomized in the MDS cohort who had a CR or PR
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 3 | 4
Months | 3.7 [3.0 to NA] — Insufficient number of participants with events | NA [0.0 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.6076, Log Rank; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: MDS Cohort: Percentage of Participants Who Achieved a Cytogenetic Response
Description: Cytogenetic response is defined as the percentage of participants who achieved a complete cytogenetic response or partial cytogenetic response according to the International Working Group (IWG) 2006 response criteria and central review. Complete cytogenetic response: Disappearance of the baseline chromosomal abnormality without appearance of new abnormalities. Partial cytogenetic response: At least 50% reduction of the chromosomal abnormality. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization up to approximately 34 months
Population: Participants randomized in the MDS cohort evaluable for cytogenetic response (ie, participants with baseline cytogenetic abnormalities).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 21 | 23
percentage of participants | 47.6 [26.26 to 68.98] | 34.8 [15.32 to 54.25]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.3840, Wald asymptotic two-sided test

6. Secondary Outcome: MDS Cohort: Kaplan-Meier Estimate of Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from randomization to the first documented progressive disease (PD), relapse, or death due to any cause during or after the treatment period, whichever occurred first, according to the International Working Group (IWG) 2006 response criteria for MDS and central review. Participants who were still alive and progression-free were censored at the date of their last response assessment. Progressive disease is defined as follows: - an increase in BM blasts relative to nadir: •If nadir less than 5% blasts: ≥ 50% increase in blasts to > 5% blasts •If nadir 5% - 10% blasts: ≥ 50% increase in blasts to > 10% blasts •If nadir 10% - 20% blasts: ≥ 50% increase in blasts to > 20% blasts •If nadir 20% - 30% blasts: ≥ 50% increase in blasts to > 30% blasts And any of the following: •At least 50% decrement from maximum remission/response levels in granulocytes or platelets •Reduction in Hgb concentration by ≥ 2 g/dL •Transfusion dependence
Time Frame: From randomization to the first documented progressive disease (PD), relapse, or death due to any cause (up to approximately 34 months)
Population: All participants randomized in the MDS cohort (PFS was a pre-specified secondary outcome measure in the MDS cohort only).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 42 | 42
Months | 8.7 [5.6 to 10.2] | 8.6 [3.4 to 11.2]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.8961, Log Rank; [statistical method as in outcome 3, analysis 1]

7. Secondary Outcome: MDS Cohort: Kaplan-Meier Estimate of Duration of Response
Description: Duration of response is defined as the time from when the first overall response (complete remission (CR), partial remission (PR), marrow complete remission (mCR), and/or hematological improvement (HI)) was observed until relapse, progressive disease (PD), or death, as defined by the International Working Group (IWG) 2006 response criteria and central review. If no relapse, PD, or death was observed, the duration of response was censored at the last response assessment date that the participant was known to be progression-free. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization to the first overall response, or death (up to approximately 34 months)
Population: Participants randomized in the MDS cohort with an overall response (CR, mCR, PR, or HI)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 26 | 20
Weeks | 33.9 [22.1 to 47.4] | 39.7 [26.3 to 73.1]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.3591, Log Rank; [statistical method as in outcome 3, analysis 1]

8. Secondary Outcome: MDS Cohort: Kaplan-Meier Estimate of Time to AML Transformation
Description: Participants were monitored for transformation to acute myeloid leukemia (AML) until death, lost to follow-up, withdrawal of consent for further data collection, or the end of the trial. Time to transformation to AML is defined as the time from the date of randomization until the date the participant had documented transformation to AML (defined as at least 30% of myeloblasts in the bone marrow). Participants with no transformation to AML were censored at the date of their last disease assessment.
Time Frame: From randomization to the date the participant had documented transformation to AML (up to approximately 34 months)
Population: All participants randomized in the MDS cohort.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 42 | 42
Months | 20.8 [15.0 to NA] — Insufficient number of participants with events | 27.7 [11.3 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.9031, Log Rank; [statistical method as in outcome 3, analysis 1]

9. Secondary Outcome: MDS Cohort: Percentage of Participants With Disease Transformation to AML
Description: Disease transformation to acute myeloid leukemia (AML) is defined as at least 30% myeloblasts in the bone marrow. Participants were monitored for transformation to AML until death, lost to follow-up, withdrawal of consent for further data collection, or the end of the trial. Participants with no transformation to AML were censored at the date of their last disease assessment.
Time Frame: From randomization until death, lost to follow-up, withdrawal of consent for further data collection, or the end of the trial (up to approximately 34 months)
Population: All participants randomized in the MDS cohort
Measure: Number; unit: Percentage of participants
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone
Number analyzed (Participants) | 42 | 42
Percentage of participants | 23.8 | 19.0

10. Secondary Outcome: AML Cohort: Kaplan Meier Estimate of Time to First Response
Description: Time to first response is defined as the time between the date of randomization and the earliest date any response (CR or CRi) was observed based on the modified International Working Group (IWG) 2003 response criteria for AML and central review. Participants who did not achieve any defined response were censored at the date of last adequate response assessment, disease progression, or death, whichever occurred first. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization and the earliest date any response (up to approximately 34 months)
Population: All participants randomized in the AML cohort
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 64 | 65
Weeks | NA [14.3 to NA] — Insufficient number of participants with events. | 25.3 [13.9 to 43.0]
Statistical Analysis 1: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.2409, Log Rank; Log-rank test stratified according to the cytogenetic risk at time of randomization (very intermediate vs poor)

11. Secondary Outcome: AML Cohort: Kaplan Meier Estimate of Relapse-free Survival
Description: Relapse-free survival is defined as time from the date of first documented response (morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi)) to the date of disease relapse or death from any cause, whichever occurred first based on the modified International Working Group (IWG) 2003 response criteria for AML and central review. Participants who were still alive and progression-free were censored at the date of their last response assessment. Participants who received a subsequent therapy before the date of disease relapse or death were censored at the time of subsequent therapy.
Time Frame: From randomization to the date of disease relapse or death from any cause, whichever occurred first (up to approximately 34 months)
Population: Participants randomized in the AML cohort with a response (CR or CRi)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 20 | 23
Months | 9.5 [5.0 to 15.0] | 12.2 [3.5 to 19.3]
Statistical Analysis 1: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.0688, Log Rank; Log-rank test stratified according to the cytogenetic risk at time of randomization (intermediate vs poor)

12. Secondary Outcome: AML Cohort: Percentage of Participants Who Achieved a Complete Cytogenetic Response
Description: Complete cytogenetic response (CyCR) based on the modified International Working Group (IWG) 2003 response criteria is defined as morphologic complete remission with a reversion to a normal karyotype. The following conditions must be met: • Absolute neutrophil count (ANC) ≥ 1.0 x10⁹/L • Platelet count ≥ 100 x10⁹/L • The bone marrow should contain less than 5% blast cells; • Auer rods should not be detectable; • No platelet, or whole blood transfusions for 7days prior to the date of the hematology assessment. AND • Reversion to normal karyotype at time of CR (based on ≥ 10 metaphases). Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization up to approximately 34 months)
Population: Participants randomized in the AML cohort evaluable for cytogenetic response (ie participants with baseline cytogenetic abnormalities).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 53 | 50
Percentage of participants | 11.3 [2.79 to 19.85] | 16.0 [5.84 to 26.16]
Statistical Analysis 1: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.4894, Wald asymptotic two-sided test

13. Secondary Outcome: AML Cohort: Percentage of Participants With Hematologic Improvement
Description: Hematological improvement was defined as participants with a erythroid response (HI-E), platelet response (HI-P) or neutrophil response (HI-NE) for at least 8 weeks, according to the IWG 2006 response criteria: Hi-E (in participants with pretreatment hemoglobin < 11 g/dL or red blood cell (RBC)-transfusion dependent): Hemoglobin increase of ≥ 1.5 g/dL, or reduction in units of RBC transfusions of at least 4 RBC transfusions/8 weeks compared with the 8 weeks prior to pretreatment. HI-P (in participants with pretreatment platelet count < 100 × 10⁹/L): Absolute increase in platelets of ≥ 30 × 10⁹/L if pretreatment value > 20 × 10⁹/L or increase from < 20 × 10⁹/L to > 20 × 10⁹/L and by at least 100%. HI-N (in participants with pretreatment neutrophils < 1.0 × 10⁹/L): At least 100% increase in neutrophils and an absolute increase of > 0.5 × 10⁹/L. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization up to approximately 34 months
Population: All participants randomized in the AML cohort (the percentage of participants with hematologic improvement was a pre-specified secondary endpoint for the AML cohort only).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 64 | 65
Percentage of participants | 42.2 [30.09 to 54.29] | 38.5 [26.63 to 50.29]

14. Secondary Outcome: AML Cohort: Kaplan-Meier Estimate of Duration of Response
Description: Duration of response is defined as the time from the first response morphologic complete remission (CR) or morphologic complete remission with incomplete blood count recovery (CRi)) was observed until relapse, PD, or death based on the IWG 2003 response criteria and central review. If no relapse, PD, or death was observed, the duration of response was censored at the last response assessment date that the participant was known to be progression-free. Response was assessed following every 3 treatment cycles until treatment discontinuation.
Time Frame: From randomization until relapse, PD, or death (up to approximately 34 months)
Population: Participants randomized in the AML cohort with an objective response (CR or CRi)
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 20 | 23
Weeks | 24.6 [16.4 to 48.0] | 52.0 [15.1 to 84.0]
Statistical Analysis 1: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.0381, Log Rank; Log-rank test stratified according to the cytogenetic risk at time of randomization (intermediate vs poor)

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse events are adverse events (AEs) that occurred or worsened on or after the first dose of study drug (durvalumab or azacitidine) and within 90 days after last dose of durvalumab or 28 days after last dose of azacitidine. A treatment-related TEAE is a TEAE where the causal relationship was assessed by the investigator as "Suspected". The intensity of AEs was graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03: Grade 1 (Mild): asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 (Moderate): minimal, local or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death due to AE.
Time Frame: From first dose to 90 days after last dose of durvalumab or 28 days after last dose of azacitidine proir to the extension study (up to approximately 34 months)
Population: All participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 38 | 41 | 64 | 62
Participants
  Any treatment-emergent adverse event (TEAE) | 38 | 41 | 64 | 62
  TEAE related to DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  TEAE related to DUR | 27 |  | 50 |
  TEAE related to AZA | 31 | 33 | 56 | 50
  TEAE related to DUR or AZA | 35 | 33 | 58 | 50
  Grade 3 TEAE | 36 | 30 | 60 | 50
  Grade 3 TEAE related to DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  Grade 3 TEAE related to DUR | 18 |  | 29 |
  Grade 3 TEAE related to AZA | 18 | 16 | 32 | 27
  Grade 3 TEAE related to DUR or AZA | 22 | 16 | 38 | 27
  Grade 4 TEAE | 33 | 27 | 43 | 34
  Grade 4 TEAE related to DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  Grade 4 TEAE related to DUR | 16 |  | 18 |
  Grade 4 TEAE related to AZA | 19 | 15 | 27 | 17
  Grade 4 TEAE related to DUR or AZA | 22 | 15 | 28 | 17
  Grade 5 TEAE | 10 | 9 | 26 | 11
  Grade 5 TEAE related to DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  Grade 5 TEAE related to DUR | 2 |  | 1 |
  Grade 5 TEAE related to AZA | 1 | 1 | 1 | 1
  Grade 5 TEAE related to DUR or AZA | 2 | 1 | 1 | 1
  Serious TEAE | 34 | 29 | 56 | 45
  Serious TEAE related to DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  Serious TEAE related to DUR | 11 |  | 33 |
  Serious TEAE related to AZA | 9 | 10 | 25 | 16
  Serious TEAE related to DUR or AZA | 14 | 10 | 34 | 16
  TEAE leading to discontinuation of DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  TEAE leading to discontinuation of DUR | 5 |  | 21 |
  TEAE leading to discontinuation of AZA | 0 | 1 | 13 | 3
  TEAE leading to discontinuation of DUR or AZA | 5 | 1 | 22 | 3
  TEAE leading to dose reduction of AZA | 3 | 6 | 10 | 2
  TEAE leading to dose interruption of DUR: number analyzed (Participants) | 38 | 0 | 64 | 0
  TEAE leading to dose interruption of DUR | 24 |  | 34 |
  TEAE leading to dose interruption of AZA | 27 | 19 | 39 | 32
  TEAE leading to dose interruption of DUR or AZA | 28 | 19 | 41 | 32
  TEAE leading to ongoing DUR infusion interruption: number analyzed (Participants) | 38 | 0 | 64 | 0
  TEAE leading to ongoing DUR infusion interruption | 2 |  | 2 |

16. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival
Description: Overall survival is defined as the time between randomization and death/censored date. Participants who were alive at the time of the clinical data cut-off were censored at the last known alive date.
Time Frame: From randomization to date of death or last known alive date (up to approximately 34 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 42 | 42 | 64 | 65
Months | 11.6 [9.5 to NA] — Insufficient number of participants with events | 16.3 [9.8 to 22.6] | 13.0 [10.3 to 17.3] | 14.4 [10.0 to 16.6]
Statistical Analysis 1: Comparison: MDS: Azacitidine + Durvalumab vs MDS: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.8973, Log Rank; [statistical method as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: AML: Azacitidine + Durvalumab vs AML: Azacitidine Alone; Test type: Other — P-values were not part of the formal testing; p = 0.0691, Log Rank; Log-rank test stratified according to the cytogenetic risk at time of randomization (intermediate vs poor)

17. Secondary Outcome: One-year Survival
Description: One-year survival is defined as the probability of survival at 1 year from randomization and is represented by the Kaplan-Meier estimate of the percentage of participants alive after 1 year.
Time Frame: At 12 months after randomization
Population: All randomized participants
Measure: Number; unit: Percentage of participants
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 42 | 42 | 64 | 65
Percentage of participants | 49 | 58 | 52 | 55

18. Secondary Outcome: Durvalumab Serum Concentration
Time Frame: Cycle 1 Day 1 end of infusion (EOI), Cycle 2 Day 1 pre-infusion, Cycle 4 Day 1 pre-infusion and EOI, and Cycle 6 Day 1 pre-infusion
Population: Participants who received at least one dose of durvalumab and who had at least 1 measurable durvalumab concentration value and with available data at each time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MDS: Azacitidine + Durvalumab | AML: Azacitidine + Durvalumab
Number analyzed (Participants) | 38 | 62
ng/mL
  Cycle 1 Day 1 end of infusion: number analyzed (Participants) | 35 | 59
  Cycle 1 Day 1 end of infusion | 375548.511 (140777.0558) | 378598.369 (201902.4363)
  Cycle 2 Day 1 pre-infusion: number analyzed (Participants) | 35 | 51
  Cycle 2 Day 1 pre-infusion | 84380.032 (92174.3455) | 54216.956 (28336.3692)
  Cycle 4 Day 1 pre-infusion: number analyzed (Participants) | 27 | 38
  Cycle 4 Day 1 pre-infusion | 132266.794 (126971.6223) | 78622.429 (41708.9956)
  Cycle 4 Day 1 end of infusion: number analyzed (Participants) | 25 | 35
  Cycle 4 Day 1 end of infusion | 433942.600 (233241.0329) | 391523.395 (147928.1261)
  Cycle 6 Day 1 pre-infusion: number analyzed (Participants) | 22 | 30
  Cycle 6 Day 1 pre-infusion | 114448.977 (64608.9007) | 142517.871 (248212.8037)

19. Secondary Outcome: Change From Baseline in Selected Hematology Parameters I
Description: Baseline values are defined as the last assessment of a particular parameter prior to administration of the participants first dose.
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 42 | 42 | 64 | 65
10^9 cells/L
  Leukocytes (10^9/L): number analyzed (Participants) | 37 | 33 | 56 | 57
  Leukocytes (10^9/L) | -1.330 (2.8158) | -0.497 (1.1452) | -2.050 (9.0236) | -0.941 (2.7708)
  Lymphocytes (10^9/L): number analyzed (Participants) | 37 | 33 | 56 | 57
  Lymphocytes (10^9/L) | -0.242 (0.5314) | -0.085 (0.3904) | -0.394 (1.6995) | -0.262 (0.9024)
  Neutrophils, Segmented (10^9/L): number analyzed (Participants) | 37 | 33 | 56 | 54
  Neutrophils, Segmented (10^9/L) | -0.665 (1.6364) | -0.266 (0.7576) | 0.646 (0.7870) | -0.102 (0.7346)
  Platelets (10^9/L): number analyzed (Participants) | 37 | 33 | 56 | 57
  Platelets (10^9/L) | 26.7 (112.92) | -2.6 (82.05) | 25.9 (92.86) | -0.9 (167.88)

20. Secondary Outcome: Change From Baseline in Selected Hematology Parameters II
Description: as for outcome 19
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 37 | 33 | 56 | 57
g/L | 2.1 (15.66) | 5.7 (18.94) | 2.2 (13.67) | -3.0 (13.91)

21. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters I
Description: as for outcome 19
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 37 | 33 | 56 | 57
g/L | -1.8 (4.01) | -1.1 (2.93) | -1.8 (5.00) | -3.8 (4.78)

22. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters II
Description: as for outcome 19
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 37 | 33 | 56 | 57
U/L
  Alkaline Phosphatase (U/L) | 8.7 (15.71) | 4.5 (13.90) | 12.3 (55.70) | 15.5 (68.53)
  Alanine Aminotransferase (U/L) | 3.6 (16.96) | 0.4 (9.40) | 0.3 (21.05) | 4.0 (19.41)
  Aspartate Aminotransferase (U/L) | 0.9 (10.52) | -0.8 (5.73) | -0.9 (16.83) | 0.5 (14.22)
  Lipase (U/L) | -5.4 (18.23) | -10.2 (25.80) | -2.0 (10.28) | 3.1 (42.85)

23. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters III
Description: as for outcome 19
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 37 | 33 | 56 | 57
mmol/L
  Calcium (mmol/L) | 0.004 (0.1013) | 0.016 (0.1008) | -0.003 (0.1523) | -0.039 (0.1189)
  Glucose (mmol/L) | -0.40 (2.210) | -0.19 (1.265) | -0.38 (2.513) | -0.02 (2.365)
  Potassium (mmol/L) | 0.15 (0.416) | -0.01 (0.451) | 0.02 (0.411) | 0.04 (0.622)
  Sodium (mmol/L) | -0.2 (2.93) | 0.3 (3.26) | -0.6 (4.49) | -1.6 (3.73)

24. Secondary Outcome: Change From Baseline in Selected Chemistry Parameters IV
Description: as for outcome 19
Time Frame: Baseline and last lab measurement collected in Cycle 2 (Last measurement could be taken either on Day 1, 8, 15 or 22)
Population: All treated participants with both non-missing baseline and postbaseline values
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
Number analyzed (Participants) | 37 | 33 | 56 | 57
umol/L
  Bilirubin (umol/L) | 2.2 (5.13) | 1.2 (4.21) | 2.4 (6.23) | -0.0 (5.31)
  Creatinine (umol/L) | -4.0 (14.77) | -2.9 (10.19) | 2.3 (16.39) | -0.6 (15.93)
  Urate (umol/L) | 6.8 (65.85) | -3.2 (67.06) | -15.1 (75.69) | -29.1 (80.85)

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from the participants first dose to their study completion (up to approximately 66 months) SAEs and Other AEs were assessed from first dose to 90 days after last dose of durvalumab or 28 days after last dose of azacitidine (up to approximately 66 months)
Arm/Group | MDS: Azacitidine + Durvalumab | MDS: Azacitidine Alone | AML: Azacitidine + Durvalumab | AML: Azacitidine Alone
All-Cause Mortality (participants affected / at risk) | 22/38 | 27/41 | 48/64 | 42/62
Serious Adverse Events (participants affected / at risk) | 34/38 | 29/41 | 56/64 | 45/62
Other Adverse Events (participants affected / at risk) | 38/38 | 40/41 | 63/64 | 60/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDS: Azacitidine + Durvalumab (N=38) | MDS: Azacitidine Alone (N=41) | AML: Azacitidine + Durvalumab (N=64) | AML: Azacitidine Alone (N=62)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 9 | 23 | 14
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 2 | 0 | 9 | 4
Generalised oedema (General disorders) | 0 | 0 | 1 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Injection site vesicles (General disorders) | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 5 | 3 | 8 | 5
Sudden death (General disorders) | 0 | 0 | 1 | 0
Cellulitis (General disorders) | 0 | 0 | 0 | 1 — Cellulitis of the right axillary region and respiratory distress
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 3 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 3 | 0
Influenza (Infections and infestations) | 1 | 1 | 3 | 0
Injection site infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Micrococcus infection (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 1 | 1 | 2
Oesophageal infection (Infections and infestations) | 0 | 1 | 0 | 0
Perineal cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 6 | 3 | 16 | 8
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 3 | 4 | 4
Septic shock (Infections and infestations) | 2 | 0 | 2 | 1
Serratia sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 2 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Superinfection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Transformation to acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 2 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 4 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDS: Azacitidine + Durvalumab (N=38) | MDS: Azacitidine Alone (N=41) | AML: Azacitidine + Durvalumab (N=64) | AML: Azacitidine Alone (N=62)
Anaemia (Blood and lymphatic system disorders) | 14 | 15 | 19 | 19
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 9
Leukopenia (Blood and lymphatic system disorders) | 8 | 3 | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 23 | 21 | 20 | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 18 | 24 | 27
Angina pectoris (Cardiac disorders) | 2 | 0 | 2 | 3
Atrial fibrillation (Cardiac disorders) | 4 | 0 | 3 | 2
Tachycardia (Cardiac disorders) | 4 | 2 | 4 | 1
Ear pain (Ear and labyrinth disorders) | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 1 | 7 | 6
Constipation (Gastrointestinal disorders) | 22 | 20 | 36 | 33
Diarrhoea (Gastrointestinal disorders) | 16 | 14 | 27 | 16
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3 | 2
Gingival bleeding (Gastrointestinal disorders) | 2 | 0 | 6 | 2
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 5 | 5
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 4
Nausea (Gastrointestinal disorders) | 16 | 11 | 26 | 22
Odynophagia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 6 | 4
Vomiting (Gastrointestinal disorders) | 10 | 10 | 20 | 15
Asthenia (General disorders) | 9 | 14 | 19 | 12
Fatigue (General disorders) | 9 | 6 | 17 | 11
General physical health deterioration (General disorders) | 0 | 3 | 1 | 1
Influenza like illness (General disorders) | 2 | 1 | 0 | 1
Injection site bruising (General disorders) | 2 | 0 | 1 | 0
Injection site erythema (General disorders) | 2 | 2 | 6 | 5
Injection site pain (General disorders) | 3 | 4 | 4 | 2
Injection site rash (General disorders) | 3 | 0 | 1 | 0
Injection site reaction (General disorders) | 3 | 4 | 10 | 7
Mucosal inflammation (General disorders) | 0 | 3 | 4 | 2
Oedema (General disorders) | 2 | 1 | 7 | 1
Oedema peripheral (General disorders) | 14 | 7 | 18 | 9
Pain (General disorders) | 3 | 1 | 1 | 2
Pyrexia (General disorders) | 12 | 13 | 23 | 21
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 3 | 1
Cellulitis (Infections and infestations) | 3 | 5 | 7 | 5
Fungal infection (Infections and infestations) | 2 | 1 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 3 | 1 | 2
Influenza (Infections and infestations) | 2 | 1 | 3 | 3
Laryngitis (Infections and infestations) | 2 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 5 | 3 | 7
Oral candidiasis (Infections and infestations) | 6 | 0 | 2 | 3
Oral herpes (Infections and infestations) | 2 | 2 | 4 | 2
Paronychia (Infections and infestations) | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 4 | 7
Tooth infection (Infections and infestations) | 2 | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 3 | 4
Urinary tract infection (Infections and infestations) | 6 | 1 | 8 | 5
Vascular device infection (Infections and infestations) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 4 | 1 | 6
Fall (Injury, poisoning and procedural complications) | 4 | 4 | 6 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 4
Alanine aminotransferase increased (Investigations) | 8 | 2 | 2 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 4 | 0 | 3 | 2
Blood bilirubin increased (Investigations) | 4 | 1 | 4 | 2
Blood creatinine increased (Investigations) | 6 | 2 | 6 | 3
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 3 | 0
Weight decreased (Investigations) | 2 | 5 | 9 | 5
Decreased appetite (Metabolism and nutrition disorders) | 8 | 7 | 18 | 10
Gout (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 3 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 2 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 0 | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2 | 13 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 4 | 5 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 3 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 5 | 4
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 11 | 7
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 15 | 6
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 8 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 12 | 3
Dizziness (Nervous system disorders) | 6 | 8 | 6 | 4
Headache (Nervous system disorders) | 8 | 3 | 6 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 4 | 3
Sciatica (Nervous system disorders) | 2 | 1 | 0 | 2
Syncope (Nervous system disorders) | 4 | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 1 | 3
Confusional state (Psychiatric disorders) | 1 | 0 | 2 | 4
Insomnia (Psychiatric disorders) | 9 | 4 | 11 | 8
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 5 | 1
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 18 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 15 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 13 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 3
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 8 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 3 | 10 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 1
Hypertension (Vascular disorders) | 2 | 2 | 4 | 4
Hypotension (Vascular disorders) | 4 | 2 | 7 | 8

LIMITATIONS AND CAVEATS:
Protocol Amendment 03 was introduced on 05 Mar 2019. At the Investigator's discretion, participants meeting all the continuation criteria were eligible to enter the optional extension phase to continue to benefit from treatment with subcutaneous azacitidine and/or durvalumab. Participants started the extension phase at the time of their next regularly scheduled dosing cycle for study drug azacitidine or azacitidine and durvalumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02775903/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02775903/SAP_001.pdf